CLINICAL TRIAL: NCT07160868
Title: Open-label Randomized Controlled Trial Investigating the Relationship Between Obstructive Sleep Apnoea and Difficult Asthma
Brief Title: Obstructive Sleep Apnoea and Difficult Asthma (OSADA)
Acronym: OSADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Tallaght University Hospital (Other)
Responsible Party: Principal Investigator, Laura Piggott, Principal Investigator, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4211
Record Dates: First submitted 2025-08-24; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Asthma (Diagnosis); OSA - Obstructive Sleep Apnea; CPAP Treatment
MeSH Terms: conditions — Asthma; Disease; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asthma - no sleep apnoea (No Intervention): This the group of asthma patients without sleep apnoea
- Asthma - sleep apnoea, no treatment (No Intervention): This the group of asthma patients with sleep apnoea (as defined as AHI ≥10 events per hour recorded) who have been randomized to the no treatment arm
- Asthma - sleep apnoea, treatment (Experimental): This the group of asthma patients with sleep apnoea (as defined as AHI ≥10 events per hour recorded) who have been randomized to the treatment arm. They will receive CPAP therapy as treatment for sleep apnoea, while monitoring their asthma control measures and airflow variability.
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Continuous positive airway pressure - device to be used at night in the treatment of sleep apnoea
  Arms: Asthma - sleep apnoea, treatment

SUMMARY:
The OSADA (Obstructive Sleep Apnoea in Difficult Asthma) trial is an open-label, randomized control trial investigating the impact of diagnosing and treating obstructive sleep apnoea (OSA) on a asthma control in patients with difficult-to-control asthma.

Participants will undergo home-based sleep studies to assess for OSA and are then allocated to one of three arms: 1) Patients with OSA treated with CPAP (intervention group), 2) Patients with OSA not treated for OSA (control group) and 3) Patients without OSA (reference group).

The primary objective is to evaluate whether treating OSA improves asthma control, symptom burden, and quality of life compared to untreated OSA and to patients without OSA. Secondary outcomes include exacerbation rates, sleep quality, and healthcare utilization.

This trial aims to clarify the contribution of OSA to poor asthma control and the potential benefits of integrated sleep and respiratory care in this complex population.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) and asthma are two of the most common respiratory disorders worldwide, with asthma estimated to affect 300 million, and OSA in the region of 1 billion people. As a result, these two disorders frequently coexist in the same person. Whilst most people with asthma achieve successful control of their condition with straightforward inhaler therapy, approximately 20% have Difficult Asthma, characterised by persistent symptoms despite high dose inhaler usage. These patients experience a significant degree of morbidity due to their asthma, with increased healthcare utilisation, limitations in activities of daily living, and an increased need for systemic corticosteroids compared to those with milder asthma. Although novel biologic therapies have improved outcomes for some of these patients, there remain significant unmet needs in the care of many.

OSA is consistently listed as an important comorbidity in Difficult Asthma, with the suggestion being that it may have a significant detrimental impact on the ability to successfully achieve asthma control. However, there is a lack of systematic assessments of the relationship between the presence and severity of OSA on asthma symptoms in Difficult Asthma cohorts, and very little is known about the effect that treating OSA has in terms of airflow variability and asthma control.

The investigators aim to conduct an open-label randomized controlled trial to study patients attending Difficult Asthma clinics. Participants will undergo home sleep studies to investigate for an underlying concurrent diagnosis of sleep apnoea. The investigators will examine baseline and longitudinal relationships between OSA and asthma exacerbations, variability of airflow (via home peak flow monitoring), patient-reported asthma control, lung function, and markers of airway inflammation over a 3-month period, allowing a comparison of patients with OSA and those without.

Patients with confirmed OSA, as defined as an apnoea-hypopnea index of ≥10 events/hour will be randomized into treatment [continuous positive airway pressure (CPAP) therapy] and no treatment groups. Again, airflow variability, exacerbation frequency, asthma control, lung function and airway inflammation will be compared between OSA patients who receive CPAP therapy and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of asthma with supportive objective diagnostics including but not limited to, variable airflow obstruction, bronchial-hyper responsiveness and demonstrable eosinophilic inflammation via fractional exhaled nitric oxide or peripheral eosinophilia
* Patients receiving step 4 or step 5 of 'The Global Initiative for Asthma' (GINA) treatment guidelines will be selected
* Between the ages of 18 to 90 years of age

Exclusion Criteria:

* Patients with previous sleep study investigations
* Excessive daytime sleepiness; ESS >17
* Previous diagnosis of a sleep disorder
* Resting hypoxaemia or need for long-term oxygen therapy
* Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in airflow variability measured by home electronic peak flow monitoring | 3-4 months
  Airflow variability will be assessed using peak expiratory flow rate (PEFR) measured with electronic home peak flow meters. Variability will be calculated using the daily amplitude percent mean (DAPM) method. Participants will be asked to record PEFR twice daily (early morning and late afternoon) over the defined period to provide adequate data points. For each day, variability will be calculated using the DAPM formula, and the average daily variability across the collection period will then be derived.

SECONDARY OUTCOMES:
Change in asthma control | 3-4 months
  As measured by;
  -Asthma Control test (ACT) scoring
Change in asthma control | 3-4 months
  As measured by;
  -Asthma quality of life questionnaire (AQLQ) score
Change in asthma control | 3-4 months
  Exacerbation frequency
Change in asthma control | 3-4 months
  Change in airway inflammation markers (FeNO)

CONTACTS AND LOCATIONS:
Locations (1):
- St. James's Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No